CLINICAL TRIAL: NCT03953547
Title: Antiplatelet Resistance Research in Patients With Peripheral Arterial Revascularization
Acronym: RAP
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RAP
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-08

CONDITIONS: Vascular Diseases
Keywords: antiplatelet resistance; peripheral arterial revascularization
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- search for antiplatelet resistance: Patients who were hospitalized in the vascular medicine department and who benefited from a search for antiplatelet resistance between April 2014 and November 2017.

SUMMARY:
In coronary pathology, persistent platelet hyperresponsiveness under antiplatelet therapy, which is often referred to as "antiplatelet resistance," is predictive of increased risk of thrombotic recurrence as well as hyper-Inhibition of this aggregation may be predictive of a hemorrhagic risk. But no study has shown that the adaptation of treatment based on platelet aggregation tests has a benefit: the management of antiplatelet treatments through the search for antiplatelet resistance (APR) is not recommended by the European Society of Cardiology (ESC) in the context of coronary angioplasty (IIIA), while this is a common practice in neurovascular pathology.

DETAILED DESCRIPTION:
In peripheral arterial disease, several studies have shown that the existence of an APR is predictive of the occurrence of thrombotic events but not all. The investigators can therefore ask the question of the benefit of adaptation of antiplatelet therapy by biological monitoring to prevent the recurrence of thrombotic events. The platelet aggregation tests used mainly concern aspirin, via stimulation with arachidonic acid, or anti-P2Y12 (clopidogrel, ticagrelor, prasugrel), via stimulation with adenosine diphosphate (ADP). For the latter, a test via the measurement of the phosphorylation of a cytoplasmic protein called "VASP" is also used routinely, making it possible to further clarify the existence of platelet resistance to anti-P2Y12. Within the vascular medicine department, any discovery of a potential resistance to the anti-platelet treatment of a patient requires a therapeutic adaptation to overcome this phenomenon of "resistance", and to improve the phenomenon of anti-aggregation

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* All patients who were hospitalized in the vascular medicine department and who received a search for antiplatelet resistance between April 2014 and November 2017.

Exclusion Criteria:

* Opposition to participation in the study
* Absence of follow-up after antiplatelet resistance testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized in the vascular medicine department and who received a search for antiplatelet resistance between April 2014 and November 2017.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of re-occlusion of the revascularization procedure | 1 year

SECONDARY OUTCOMES:
Number of cardiovascular events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël ATTAL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Siller-Matula JM, Delle-Karth G, Lang IM, Neunteufl T, Kozinski M, Kubica J, Maurer G, Linkowska K, Grzybowski T, Huber K, Jilma B. Phenotyping vs. genotyping for prediction of clopidogrel efficacy and safety: the PEGASUS-PCI study. J Thromb Haemost. 2012 Apr;10(4):529-42. doi: 10.1111/j.1538-7836.2012.04639.x. PMID 22260716
- [Result] Pinto Slottow TL, Bonello L, Gavini R, Beauzile P, Sushinsky SJ, Scheinowitz M, Kaneshige K, Xue Z, Torguson R, Tantry U, Pichard AD, Satler LF, Suddath WO, Kent K, Gurbel P, Waksman R. Prevalence of aspirin and clopidogrel resistance among patients with and without drug-eluting stent thrombosis. Am J Cardiol. 2009 Aug 15;104(4):525-30. doi: 10.1016/j.amjcard.2009.04.015. Epub 2009 Jun 24. PMID 19660606
- [Result] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Result] Gupta R, Moore JM, Griessenauer CJ, Adeeb N, Patel AS, Youn R, Poliskey K, Thomas AJ, Ogilvy CS. Assessment of Dual-Antiplatelet Regimen for Pipeline Embolization Device Placement: A Survey of Major Academic Neurovascular Centers in the United States. World Neurosurg. 2016 Dec;96:285-292. doi: 10.1016/j.wneu.2016.09.013. Epub 2016 Sep 15. PMID 27641263
- [Result] Mazur P, Frolow M, Nizankowski R, Sadowski J, Undas A. Impaired responsiveness to clopidogrel and aspirin in patients with recurrent stent thrombosis following percutaneous intervention for peripheral artery disease. Platelets. 2013;24(2):151-5. doi: 10.3109/09537104.2012.676220. Epub 2012 Apr 13. PMID 22497730
- [Result] Mueller MR, Salat A, Stangl P, Murabito M, Pulaki S, Boehm D, Koppensteiner R, Ergun E, Mittlboeck M, Schreiner W, Losert U, Wolner E. Variable platelet response to low-dose ASA and the risk of limb deterioration in patients submitted to peripheral arterial angioplasty. Thromb Haemost. 1997 Sep;78(3):1003-7. PMID 9308744
- [Result] Kasotakis G, Pipinos II, Lynch TG. Current evidence and clinical implications of aspirin resistance. J Vasc Surg. 2009 Dec;50(6):1500-10. doi: 10.1016/j.jvs.2009.06.023. Epub 2009 Aug 12. PMID 19679423
- [Result] Doly JS, Lorian E, Desormais I, Constans J, Bura Riviere A, Lacroix P. [Prevalence and prognosis of aspirin resistance in critical limb ischemia patients]. J Mal Vasc. 2016 Dec;41(6):358-364. doi: 10.1016/j.jmv.2016.08.004. Epub 2016 Oct 14. French. PMID 27745943
- [Result] Navarese EP, Wernly B, Lichtenauer M, Petrescu AM, Kolodziejczak M, Lauten A, Frediani L, Veulemanns V, Wanha W, Wojakowski W, Lesiak M, Ferrante G, Zeus T, Tantry U, Bliden K, Buffon A, Contegiacomo G, Jung C, Kubica J, Pestrichella V, Gurbel PA. Dual vs single antiplatelet therapy in patients with lower extremity peripheral artery disease - A meta-analysis. Int J Cardiol. 2018 Oct 15;269:292-297. doi: 10.1016/j.ijcard.2018.07.009. Epub 2018 Jul 3. PMID 30045826
- [Result] Soden PA, Zettervall SL, Ultee KH, Landon BE, O'Malley AJ, Goodney PP, DeMartino RR, Arya S, Schermerhorn ML; Society for Vascular Surgery Vascular Quality Initiative. Dual antiplatelet therapy is associated with prolonged survival after lower extremity revascularization. J Vasc Surg. 2016 Dec;64(6):1633-1644.e1. doi: 10.1016/j.jvs.2016.05.098. Epub 2016 Aug 27. PMID 27575814